CLINICAL TRIAL: NCT04767698
Title: Addition of Belimumab to B-cell Depletion to Produce Prolonged Remission of Relapsing-remitting Multiple Sclerosis Disease Activity
Brief Title: Addition of Belimumab to B-cell Depletion in Relapsing-remitting Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding source decided to stop funding the study.
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00246563
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belimumab + short-term Ocrelizumab (Experimental): Participants will receive Belimumab and Ocrelizumab.
  Interventions: Drug: Belimumab; Drug: Short-course Ocrelizumab
- Continued Ocrelizumab (Active Comparator): Participants will receive Ocrelizumab only.
  Interventions: Drug: Continued Ocrelizumab

INTERVENTIONS:
Drug: Belimumab — 200 mg SC weekly for 36 months
  Arms: Belimumab + short-term Ocrelizumab
Drug: Short-course Ocrelizumab — 300 mg, two infusions two weeks apart and then 600 mg as a single infusion after six months (only one time) (total of two courses of treatment)
  Arms: Belimumab + short-term Ocrelizumab
Drug: Continued Ocrelizumab — 300 mg, two infusions two weeks apart and then 600 mg as a single infusion every six months for a total of 36 months
  Arms: Continued Ocrelizumab

SUMMARY:
Multiple sclerosis is the most common inflammatory disease of the central nervous system and a common cause of disability in young adults. Depleting B cells from the circulation with an anti-cluster of differentiation (CD) 20 antibodies has proven to be an effective strategy in reducing relapses and disability in patients with the relapsing-remitting disease. However, continuous and long-term depletion of B-cells can result in reduced immunoglobulin levels, immunosuppression, and an increased tendency for severe infections and perhaps, even malignancy.

Blocking B-cell Activating Factor (BAFF) is effective for the treatment of several autoimmune disorders. Belimumab, a BAFF blocking antibody, has been approved by the Food and Drug Administration for the treatment of systemic lupus erythematosus. Belimumab has been shown to have immunomodulatory properties, without resulting in overt immunosuppression.

The investigators hypothesize that belimumab, given to patients who received a short course of treatment with B-cell depleting antibody (ocrelizumab), will be safe and equally effective in reducing MS disease activity (as compared to patients receiving continuous treatment with ocrelizumab); while resulting in less immunosuppression, as measured by antibody response to pneumococcal vaccination. Currently, available treatment strategies in relapsing MS sacrifice higher efficacy for long-term safety or vice versa. The proposed strategy in this application combines the long-term safety and high efficacy to treat patients with relapsing-remitting multiple sclerosis (RRMS) and, if eventually proven effective, can be adopted in a large proportion of patients with this chronic disease.

This is a randomized, open-labeled trial. Forty eligible participants will be randomized 1:1 to either receiving a form of standard of care, ocrelizumab (300 mg two infusions two weeks apart at baseline and then 600 mg as a single infusion every six months) or belimumab (200 mg subcutaneous (SC) weekly for 36 months) plus two courses of ocrelizumab (300 mg two infusions two weeks apart at baseline and 600 mg as a single infusion six months later). Co-primary outcomes of the study include pneumococcal vaccine antibody response, the return of MS disease activity, and proportions of patients with adverse events and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS based on McDonald criteria 2017
* Age > 18
* A clinical relapse in the past 12 months OR an enhancing lesion on brain/ spinal cord MRI in the past 6 months OR a new T2/FLAIR lesion on a brain/spinal cord MRI obtained in the past 6 months (compared to a previous MRI obtained within one year from the latest MRI)
* Pre-existing pneumococcal antibody titers (>1.0 mg/mL) to =<9 of 23 vaccine serotypes
* Female Subjects: Not pregnant or nursing and at least one of the following conditions apply: a. Non- childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea. b. Child-bearing potential and agrees to use one of the contraception methods as described by the investigator or designee, from Day 0 until 24 weeks after the last dose of study medications (See details below).
* Liver function at the time of screening: alanine aminotransferase (ALT) < 2x upper limit of normal (ULN); bilirubin <= 1.5x ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Prior therapy at any time: has ever received any of the following: a) B-cell targeted therapy (e.g., rituximab, ocrelizumab, other anti-cluster of differentiation (CD)20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], B lymphocyte stimulator (BLyS)-receptor fusion protein [BR3], Transmembrane activator and calcium-modulating ligand (CAML) interaction (TACI) fragment, crystallizable (Fc), or belimumab)
* Prior use of cladribine, mitoxantrone, cyclophosphamide, or hematopoietic stem cell transplantation (HSCT)
* Lymphopenia: a lymphocyte count <500/ millimeter (mm)^3
* Neutrophils <1.5x 10E9/L.
* Drug sensitivity: a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergies including a previous anaphylactic reaction to parenteral administration contrast agents, human or murine proteins or monoclonal antibodies
* Treatment with steroids in the last 30 days
* Clinically unstable medical or psychiatric disorder
* Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, poses a significant suicide risk
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies
* Substance abuse: has evidence of current drug or alcohol abuse or dependence
* 365 Day prior therapy: has received a biologic investigational agent other than B-cell targeted therapy [e.g., abetimus sodium, anti CD40L antibody (e.g., BG9588/ IDEC-131; investigational agent applies to any drug not approved for sale in the country in which it is being used]
* 30 Day prior therapy: has received any of the following within 30 days before Day 0: a) Any other MS disease-modifying therapy, not mentioned above (including fumaric acid esters, sphingosine-1-phosphate (S1P) receptor modulators, teriflunomide, and natalizumab). Glatiramer acetate and interferons are permitted up to the day of starting the investigational medication. Intravenous, oral, and Inhaled steroids and new topical immunosuppressive agents (e.g., eye drops, topical creams) are allowed.
* 30 Day prior therapy: has received a live virus vaccine or a non-biologic investigational agent.
* Malignancy: has a history of malignancy in the past 5 years except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Have a history of a primary immunodeficiency
* Have a significant IgG deficiency (IgG level < 400 mg/dL)
* Have an IgA deficiency (IgA level < 10 mg/dL)
* Infection history:

  * Currently on any suppressive therapy for chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria)
  * Hospitalization for treatment of infection within 60 days of Day 0.
  * Use of parenteral (IV or IM) antibiotics (anti-bacterial, antiviral, anti-fungal, or anti-parasitic agents) within 60 days of Day 0
* Other disease/conditions: has any of the following: a) clinical evidence of significant unstable or uncontrolled acute or chronic diseases (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk; b) a surgical procedure planned in the 6 months after Day 0; c) a known history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the investigator, makes the subject unsuitable for the study
* Hepatitis status:

  * Serologic evidence of current or past Hepatitis B (HB) infection based on the results of testing for HBsAg and HBcAb as follows: Patients positive for HBsAg or HBcAb are excluded
  * A positive test for Hepatitis C antibody
* HIV: known to have a historically positive HIV test or tests positive at screening for HIV.
* Laboratory abnormalities: has an abnormal laboratory assessment, which is judged clinically significant by the investigator.
* Drug Sensitivity: has a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergies including a previous anaphylactic reaction to parenteral administration contrast agents, human or murine proteins or monoclonal antibodies that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Any contraindication to undergoing MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Bhargava, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One (1) participant did not meet one of the inclusion criteria (pre-existing pneumococcal antibody titers to =<9 of 23 vaccine serotypes) during screening and was therefore excluded.
Groups:
- Belimumab + Short-term Ocrelizumab: Participants will receive Belimumab and Ocrelizumab.
  Belimumab: 200 mg subcutaneous (SC) weekly for 36 months
  Short-course Ocrelizumab: 300 mg, two infusions two weeks apart and then 600 mg as a single infusion after six months (only one time) (total of two courses of treatment)
Period: Overall Study
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Started | 1 | 2
Completed (Study was terminated) | 0 | 0
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: No data was collected because the trial was prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pneumococcal Vaccine Antibody Response
Description: The proportion of patients with positive antibody responses to >/=1 of the 23 pneumococcal vaccine serotypes measured four weeks post-vaccination (vaccination given at month 24). A positive antibody response is defined as a two-fold increase from pre-vaccination levels against >/=1 of the 23 pneumococcal serotypes measured.
Time Frame: Month 25
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Safety as Assessed by Adverse Events
Description: Adverse events (AEs) and serious adverse events (SAEs), including AEs of special interest (opportunistic infections, herpes zoster, malignancies, hypersensitivity and infusion reactions, suicidal ideation, intent or behavior and all-cause mortality).
Time Frame: 24 months
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Difference Between the Two Treatment Groups in GM-CSF/IL-10 Ratio
Description: Granulocyte-macrophage colony-stimulating factor (GM-CSF)/Interleukin (IL)-10 ratio (produced by stimulated repopulated B-cells).
Time Frame: Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Difference Between the Two Treatment Groups in IL-6/IL-10 Ratio
Description: IL-6/IL-10 ratio (produced by stimulated repopulated B-cells).
Time Frame: Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Assessment of Return of Disease Activity by Month 24
Description: Proportions of patients with a return of the disease activity, as objectively demonstrated by the development of new T2 hyperintense lesions or Gd-enhancing lesions on the MRI (noted on a scan performed more than six months after treatment initiation) or a clinical relapse, defined as new or worsening neurologic symptom(s) with an objective change on the EDSS of at least 1.5 points for participants with baseline EDSS scores of 0 or 0.5 and at least 1-point change for participants with EDSS of 1 or more, as determined by the examining neurologist. Symptoms must have been attributable to multiple sclerosis (MS), last ≥48 hours, been present at normal body temperature, and preceded by at least 30 days of clinical stability.
Time Frame: Month 24
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Assessment of Return of Disease Activity by Month 36
Description: Proportions of patients with a return of the disease activity, as objectively demonstrated by the development of new T2 hyperintense lesions or Gd-enhancing lesions on the MRI (noted on a scan performed more than six months after treatment initiation) or a clinical relapse, defined as new or worsening neurologic symptom(s) with an objective change on the EDSS of at least 1.5 points for participants with baseline EDSS scores of 0 or 0.5 and at least 1-point change for participants with EDSS of 1 or more, as determined by the examining neurologist. Symptoms must have been attributable to MS, last ≥48 hours, been present at normal body temperature, and preceded by at least 30 days of clinical stability.
Time Frame: Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Assessment of Clinical Disease Activity by Month 24
Description: Annualized relapse rate (ARR) which is the number of relapses divided by the number of follow up years.
Time Frame: Month 24
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Assessment of Clinical Disease Activity by Month 36
Description: Annualized relapse rate (ARR) which is the number of relapses divided by the number of follow up years.
Time Frame: Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Proportion of Participants With a Three-month Confirmed Increase in EDSS Score
Description: Assessment of disability progression by the proportion of participants with a three-month confirmed increase in Expanded Disability Status Scale (EDSS) score.
Time Frame: Month 24
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Proportion of Participants With a Three-month Confirmed Increase in EDSS Score
Description: as for outcome 9
Time Frame: Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Proportion of Participants With a Three-month Confirmed Decrease in EDSS Score
Description: Assessment of disability progression by the proportion of participants with a three-month confirmed decrease in EDSS score.
Time Frame: Month 24
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Proportion of Participants With a Three-month Confirmed Decrease in EDSS Score
Description: as for outcome 11
Time Frame: Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Serum Neurofilament Light Chain (NfL) in pg/mL
Description: Assessment of a serum biomarker of neuroaxonal degeneration.
Time Frame: Baseline and Month 24
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Serum Neurofilament Light Chain (NfL) in pg/mL
Description: Assessment of a serum biomarker of neuroaxonal degeneration.
Time Frame: Baseline and Month 36
Population: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No data was collected
Description: No data was collected
Arm/Group | Belimumab + Short-term Ocrelizumab | Continued Ocrelizumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was prematurely terminated and therefore there was no data collected nor analysis performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04767698/Prot_SAP_000.pdf